CLINICAL TRIAL: NCT01254058
Title: Novel Vision Testing Paradigms for Patients With Glaucoma
Brief Title: Saccadic Eye Movements Are Impaired In Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB 06-056
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma Group
- Age-Matched Controls

SUMMARY:
The purpose of this study is to determine whether rapid eye movements called saccades are impaired in glaucoma, a neurodegenerative disease of visual pathways.

DETAILED DESCRIPTION:
Eye movements that quickly scan a visual scene are critical to a number of daily activities including driving. It is not known whether rapid eye movement called saccades, are altered in glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Ages from 40-80 years. Primary open angle glaucoma is defined by characteristic glaucomatous optic nerve head findings and the presence of corresponding visual field deficits in one or both eyes. All control subjects will be age-matched, with no ocular medical or surgical history, and a completely normal eye examination. Age-matched controls will be recruited from local hospital personnel and accompanying relatives.

Exclusion criteria:

* Any patient with a history of other eye disease, neurological disease or neurodegenerative disorder, or history of incisional ocular surgery within the previous month will be excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 19 glaucoma patients and 21 age-matched controls will be identified and consented.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Delay in saccades | April 2014

CONTACTS AND LOCATIONS:
Overall Officials: Neeru Gupta, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Gupta N, Krishnadev N, Hamstra SJ, Yucel YH. Depth perception deficits in glaucoma suspects. Br J Ophthalmol. 2006 Aug;90(8):979-81. doi: 10.1136/bjo.2006.091025. Epub 2006 May 3. PMID 16672326
- [Result] Kanjee R, Yucel YH, Steinbach MJ, Gonzalez EG, Gupta N. Delayed saccadic eye movements in glaucoma. Eye Brain. 2012 Nov 26;4:63-68. doi: 10.2147/EB.S38467. eCollection 2012. PMID 28539782